CLINICAL TRIAL: NCT02350530
Title: A Phase II Study to Evaluate the Surgical Conversion Rate in Patients With RAS Mutation-type Receiving FOLFOXIRI +/- Bevacizumab for Unresectable Colorectal Liver-Limited Metastases
Brief Title: FOLFOXIRI With or Without Bevacizumab as First-line Treatment for Unresectable Liver-only Metastatic Colorectal Cancer Patients With RAS Mutation-type
Acronym: FORBES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Associate professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU09
Record Dates: First submitted 2015-01-24; First posted 2015-01-29 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Metastatic colorectal cancer; Liver metastases; Liver resection; Liver ablation; Conversion therapy; FOLFOXIRI; Oxaliplatin; Irinotecan; Fluorouracil; Bevacizumab; RAS mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Oxaliplatin; Fluorouracil; FOLFOXIRI protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (FOLFOXIRI + Bevacizumab) (Experimental): FOLFOXIRI + Bevacizumab
  Interventions: Drug: FOLFOXIRI + Bevacizumab
- B (FOLFOXIRI) (Active Comparator): FOLFOXIRI
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI + Bevacizumab — Bevacizumab 5mg/kg + irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle until PD or resectability or to max. 12 cycles
  Other Names: Bevacizumab; Irinotecan; Oxaliplatin; 5-Fluorouracil
  Arms: A (FOLFOXIRI + Bevacizumab)
Drug: FOLFOXIRI — Irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle until PD or resectability or to max. 12 cycles
  Other Names: Irinotecan; Oxaliplatin; 5-Fluorouracil
  Arms: B (FOLFOXIRI)

SUMMARY:
BACKGROUND:

For patients with liver-limited metastatic colorectal cancer (mCRC), complete resection of liver metastases is the only potentially curative treatment. The current goal of medical treatment for colorectal cancer with initially unresectable liver metastases is to maximize the rate of secondary resection and prolong overall survival (OS). A strong correlation was found between response rate and secondary resection rate of metastases, and the triple drugs combination of infusional 5-fluorouracil/leucovorin (5-FU/LV), irinotecan, and oxaliplatin (FOLFOXIRI) was recommended can be used in selected patients with potentially resectable metastases in order to improve response rate and make resection more possible. The addition of a anti-VEGFs monoclonal antibody such as bevacizumab to chemotherapy has been shown to increase response rate, resection rate and improve OS in the first-line treatment of mCRC patients. The efficacy and safety of bevacizumab in addition to triplet drugs were previously tested in OLIVIA trial, the resection rate of liver metastases of 49% was reported, and the response rate was 81%; most common grade 3-4 adverse events was neutropenia. On the basis of such promising results, we conducted the present randomized study to explore whether FOLFOXIRI plus bevacizumab compared with FOLFOXIRI alone as first-line treatment could improve radical resectability in patients with RAS mutation-type, unresectable liver-only metastatic colorectal cancer.

OBJECTIVE:

The primary objective of the FOBULM study is to evaluate the efficacy of FOLFOXIRI plus bevacizumab compared to FOLFOXIRI alone in patients with initially unresectable liver-limited RAS mutation-type mCRC.

Secondary objectives are safety and tolerability of the treatment, efficacy in terms of objective response rate (ORR), OS, progression free survival (PFS), quality of life and an assessment of biomarkers for predictive response and prognosis.

DETAILED DESCRIPTION:
OVERVIEW OF TRIAL DESIGN

This FOCULM trial is a a two-arm, multicenter, open labelled, prospective, randomized phase II studies. Eligible patients with initially unresectable liver-limited mCRC will be randomised 1:1 to receive either FOLFOXIRI plus bevacizumab or FOLFOXIRI alone.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum.
3. Male or female subjects > 18 years < 70 of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. There must be documentation by CT scan, MRI, or intraoperative palpation that the patient has evidence of metastases confined to the liver.
6. The liver metastases must have been assessed by multidisciplinary team including hepatic surgeon approved to participate in the study to be unresectable based on at least one of the four criteria: 1. All of the liver metastases can not be completed resected with negative margins; 2. No ability to preservation of two contiguous hepatic segments; 3. No ability to preservation of adequate vascular inflow and outflow as well as biliary drainage; 4. Complete resection would require greater than 70% of the liver parenchyma to be removed.
7. The colorectal primary tumor or metastatic tumor must be determined to be KRAS (exon 2 at codon 12 and 13; exon 3 at codon 59 and 61; exon 4 at codon 117 and 146) or NRAS (exon 2 at codon 12 and 13; exon 3 at codon 59 and 61; exon 4 at codon 117 and 146) mutation-type.
8. Primary tumor and regional nodes were resected with clear surgical margins or; unresected primary tumor with plan to radical resect the primary tumor.
9. No previous any systemic anticancer therapy for metastatic disease (adjuvant chemotherapy for non-metastatic disease is allowed if terminated more than 6 months ago).
10. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment: Hemoglobin (Hb) ≥ 90g/ L, absolute neutrophil count (ANC) ≥ 1.5×109/ L, platelet count ≥ 100×109/ L; Total bilirubin ≤ 1.5×the upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 ×ULN; Serum creatinine ≤1.5×the ULN.

Exclusion Criteria:

1. Any evidence of extrahepatic metastases, lymph node (including portal lymph nodes) metastases and primary tumor recurrence.
2. Previous hepatic resection and/or ablation, hepatic arterial infusion therapy, radiation therapy to the liver.
3. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization.
4. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
5. Heart failure grade III/IV (NYHA-classification).
6. Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.
7. Subjects with known allergy to the study drugs or to any of its excipients.
8. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
9. Breast- feeding or pregnant women
10. Lack of effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The conversion rate of liver metastases | 8 months
  Defined as the proportion of patients who had a curative liver treatment following protocol treatment, i.e., liver metastases that can be radical resected with or without ablation with no postoperative evidence of residual malignant disease.

SECONDARY OUTCOMES:
Toxicity assessed using the NCI common toxicity criteria, version 4.0. | 8 months
  The grade of toxicity will be assessed using the NCI common toxicity criteria, version 4.0.
Response rate | 8 months
  CR + PR rate will be assessed according to the RECIST version 1.1 guidelines.
Overall survival time | 5 years
  Estimated from the date of randomization to death from any cause.
Progression free survival | 2 years
  Time measured from the day of randomization to the date of first documented progression, or death from any cause.
Quality of life (QLQ C30) | Every 2 weeks after the first treatment until 6 months
  Scores according to EORTC QLQ-C30 scoring manual

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, M.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China